CLINICAL TRIAL: NCT06933420
Title: Feasibility/First in Human Study of Visible Spectrum, Low Level, Microbicidal Light-based Intravaginal Therapy for Treatment of Yeast and Bacterial Vaginitis
Brief Title: Clinical Protocol CERN Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cern Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CERN-PR-001
Record Dates: First submitted 2025-03-21; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Bacterial Vaginosis; Fungal Vaginal Infections
MeSH Terms: conditions — Vaginosis, Bacterial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bacterial Vaginosis and Fungal Vaginitis (Experimental): For bacterial vaginosis, the participants receive 30-minute daily treatment with the Cern Device for 5 days. For fungal vaginitis, the participants receive 60-minute daily treatment with the Cern Device for 5 days.
  Interventions: Device: Cern Device

INTERVENTIONS:
Device: Cern Device — The Cern Device is an Intravaginal device utilizing low level microbicidal visible light at a 450nm low level microbicidal light, in visible spectrum for treatment of vaginitis, including both bacterial vaginosis and fungal vaginitis.

SUMMARY:
The goal of this clinical trial is to learn if the intravaginal Cern device works to treat bacterial vaginosis and fungal vaginitis in premenopausal women. It will also learn about the safety of the device. The main questions it aims to answer are: Does the device accomplish symptom resolution and negative diagnostic tests post-treatment? What medical problems do participants have when using the intravaginal device? Participants will use the investigational intravaginal device for 5 consecutive days, participate in teleconferences and weekly follow-ups, attend in-clinic visits, and maintain a study diary.

DETAILED DESCRIPTION:
The CERN Feasibility Study is an interventional clinical trial designed to evaluate the Cern Medical Device in the treatment of bacterial vaginosis and fungal vaginitis. The study assesses both the efficacy and safety of this innovative technology, which combines 450nm visible spectrum light with a natural photosensitizer (carboxy methyl cellulose and curcumin). The primary objective is to determine the device's effectiveness by measuring symptom resolution and negative diagnostic tests post-treatment. The secondary objective focuses on safety, monitoring adverse effects and patient tolerance during and after treatment. The study design involves recruiting up to 30 premenopausal women with culture-confirmed bacterial vaginosis or fungal vaginitis. Participants are divided into two groups, in the bacterial vaginosis group, the device is used for 30 minutes daily for 5 consecutive days. And in the fungal vaginitis group, the device is used for 60 minutes daily for 5 consecutive days. Following treatment, participants undergo a 45-day follow-up period, which includes daily telecom check-ins during treatment, weekly follow-ups, and a final assessment at 28 days post-treatment. Adherence is tracked through daily diaries and telecom follow-ups, ensuring treatment compliance, effectiveness monitoring, and adverse reaction tracking. Treatment success is determined by self-reported symptom resolution and negative diagnostic cultures, while safety is assessed through self-reported adverse events and clinical examinations.

ELIGIBILITY:
Inclusion Criteria:

* Confirm symptomatic and laboratory-confirmed bacterial vaginosis or fungal vaginitis

Exclusion Criteria:

* Postmenopausal status, current use of intravaginal devices, concurrent medical therapy for fungal vaginitis or bacterial vaginosis, recent medical therapy for vaginitis in past 7 days, immunosuppressive medication ≤ 3 months before screening, radiation therapy ≤ 3 months before screening, known allergy to curcumin, acrylic, or silicone, major organ disease or clinically significant infection or conditions that may affect clinical assessment of vaginitis, pregnancy or plans for pregnancy, history of intolerance to intravaginal devices, symptomatic pelvic organ prolapse stage 2 or greater.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Premenopausal women
Enrollment: 9 (Estimated)
Dates: Start 2024-11-06 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Resolution of Clinical Symptoms | Day 1 to Day 28 (post-treatment)
  Number of participants reporting resolution of vaginal discharge, itching, burning, and/or irritation, assessed using a symptom severity scale with the following levels: none, mild, moderate, or severe. Improvement is defined as a reduction in symptom severity to "none" or "mild" for all reported symptoms.
Negative Diagnostic Test Result | Within 7 days after treatment completion
  Number of participants with a negative laboratory test for bacterial vaginosis or fungal vaginitis.

SECONDARY OUTCOMES:
Safety of the Cern Device | Day 1 to Day 45
  Number of participants reporting any device-related adverse events (e.g., discomfort, irritation, pain) during or after use of the device. Events will be captured via daily treatment diaries, daily telehealth check-ins, and post-treatment follow-up calls.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Akerman Med, Irvine, California
  - Akerman Med, Orange, California
  - Akerman Med, Santa Ana, California